CLINICAL TRIAL: NCT05462652
Title: Project STAND (Self-guided Treatment for Adolescents Navigating Depression): a Randomized Controlled Trial
Brief Title: Self-guided Treatment for Adolescents Navigating Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Limbix Health, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LMX-001
Record Dates: First submitted 2022-07-14; First posted 2022-07-18 (Actual); Results first posted 2024-06-12 (Actual); Last update posted 2024-06-12 (Actual); Status verified 2024-05

CONDITIONS: Depressive Symptoms; Depression; Depressive Disorder; Depressive Episode
Keywords: Mental Health; Adolescents; Depression; Adolescent Mental Health
MeSH Terms: conditions — Depression; Depressive Disorder; Psychological Well-Being

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Active Intervention (Experimental): The active intervention is a 5-week program divided into 5 levels intended to be completed weekly. Each level is expected to take about 60 minutes to complete. Activities in each level may include reading text on the screen, answering multiple choice style questions, swiping or clicking a button to move through screens, dragging and dropping elements on screen, and completing tasks outside of the app. Certain on-demand resources can be accessed in the apps at any time, including crisis resources. Where appropriate, text entries in the app that match a database of concerning words/phrases will trigger an automated pop-up suggesting participants visit the in-app crisis resources if they need additional support. Text entries will also be monitored by study staff for safety, though not in real-time. Participants will be instructed to complete a weekly PHQ-8 assessment in the mobile app.
  Interventions: Device: Active Intervention
- Usual Care (No Intervention): UC is based on a stepped care model for treatment for symptoms of depression. It can include any of the following: active monitoring of depressive symptoms and suicidality, supportive counseling by a healthcare provider, psychosocial support interventions, collaborative care (e.g. facilitation of parental and patient self-management, referral for peer support or other community or school-based behavioral health programs), psychoeducation, complementary and alternative medicine approaches, psychotherapy (e.g. behavioral treatment, interpersonal therapy, cognitive behavioral therapy), pharmacotherapy for mood problems, visit to a primary care provider, behavioral or mental health specialist or therapist, counselor or coach for mood disorder. For purposes of this study, UC will be enhanced by prompting participants to complete a weekly PHQ-8 assessment in a mobile app.

INTERVENTIONS:
Device: Active Intervention — The active intervention is a 5-week program divided into 5 levels intended to be completed weekly. Each level is expected to take about 60 minutes to complete. Activities in each level may include reading text on the screen, answering multiple choice style questions, swiping or clicking a button to move through screens, dragging and dropping elements on screen, and completing tasks outside of the app. Certain on-demand resources can be accessed in the apps at any time, including crisis resources. Where appropriate, text entries in the app that match a database of concerning words/phrases will trigger an automated pop-up suggesting participants visit the in-app crisis resources if they need additional support. Text entries will also be monitored by study staff for safety, though not in real-time. Participants will be instructed to complete a weekly PHQ-8 assessment in the mobile app.
  Arms: Active Intervention

SUMMARY:
The goal of this study is to test whether an investigational mobile app can be a helpful treatment option for adolescents with symptoms of depression. Adolescents aged 13 to 21 with depression symptoms can be part of this study if eligible.

Eligible participants will be randomly assigned to one of two groups: one group will receive the mobile app intervention in addition to their usual care and the other group will simply continue their usual care for symptoms of depression. Both groups will have 5 weeks to use a study app, and will complete assessments during the intervention period, at post-intervention, and at one month follow-up.

DETAILED DESCRIPTION:
The primary aim of the proposed research is to evaluate the effectiveness of a self-guided, cognitive behavioral therapy (CBT)-based mobile app + assessment-enhanced Usual Care (eUC) compared to eUC alone as an intervention for adolescents with symptoms of depression who are under the supervision of a licensed healthcare provider.

The sample size for this study is 220 subjects. Sample size calculation is based on primary outcome patient health questionnaire (PHQ-8) at post-intervention (5 weeks). Six PHQ-8 measurements will be collected from each subject (baseline and weekly during the 5-week intervention period). Using a two-sample t-test approach, assuming a two-tailed alpha set at 0.05, a total of 200 participants (100 in each study arm) will give us 80% power to detect a moderate effect size of at least d=0.4. Given an anticipated 10% rate of attrition, we aim to enroll 220 total participants in the study.

A 50% female sample will be targeted. Earlier recruitment efforts within the study demographic have resulted in majority female samples, consistent with prevalence rates within the study population. As such, recruitment efforts will be undertaken to ensure representation of male participants. Recruitment efforts will be taken to ensure adequate representation of underrepresented racial and ethnic minority groups.

Children between the ages of 13-17 will be included in this research as the program to be evaluated is specifically designed as an intervention for adolescents with symptoms of depression. Assent will be obtained from all children under 18 for study enrollment unless legally emancipated or financially independent in accordance with CA state regulations and regulations of the state in which the minor resides.

Study staff will monitor participants' symptom deterioration and questionnaire data for safety.

ELIGIBILITY:
Inclusion Criteria:

* 13-21 years of age
* PHQ-8 score ≥ 5 at eligibility screening
* English fluency and literacy (participant and legal guardian, if applicable)
* Access to a compatible smartphone (or other device) and operating system (i.e., capable of installing the app from the Google Play or Apple App Store; list will be provided on study website) and regular internet access
* Participant willing and able to provide informed consent/assent and have legal guardian willing and able to provide informed consent (if required)
* Under the care of a United States (U.S.)-based licensed healthcare provider and willing to provide contact information for the provider and sign a HIPAA release that allows Limbix to contact provider
* Willing and able to provide information required for study enrollment (e.g. all responses to initial PHQ-8 assessment, and current antidepressant medication status)
* Located in the continental U.S., Hawaii, or Alaska, and not planning to leave the U.S. during the study period (through 1-month follow up assessments, up to 11 weeks after eligibility screening)

Exclusion Criteria:

* Diagnosis of (or treatment for) bipolar disorder, post traumatic stress disorder, psychotic disorder, substance use disorder, or eating disorder within the 12 months prior to eligibility screening
* Change in psychotropic medication (initiation or change in dose) within the 30 days prior to eligibility screening
* Plans to initiate or change treatment (e.g., psychotherapy, psychotropic medication, and/or other psychosocial treatment) for a mental health disorder during the study intervention period (5 weeks) as determined at eligibility screening
* Suicide attempt within the past year
* Active suicide ideation with intent
* Previous participation in user testing or clinical testing of Spark or SparkRx, or other previous use of SparkRx app
* Participation in any other clinical research involving a mental health intervention or treatment within 60 days prior to eligibility screening
* Plans to participate in any other clinical research involving a mental health intervention or treatment during the study intervention period (5 weeks) as determined at eligibility screening
* Any condition, comorbidity, or event that, in the opinion of the investigator, will prevent the participant from adhering to the protocol or benefitting from the intervention or will prevent investigators from being able to ensure safety
* Having a sibling who is a past or current participant in the study

Ages: 13 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 223 (Actual)
Dates: Start 2022-07-28 (Actual); Primary Completion 2023-04-21 (Actual); Study Completion 2023-04-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aarthi Padmanabhan, PhD, Principal Investigator — Limbix Health, Inc.
Locations (1):
- Limbix Health, Inc., San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Furman DJ, Hall SA, Avina C, Kulikov VN, Lake JI, Padmanabhan A. Assessing the Efficacy and Safety of a Digital Therapeutic for Symptoms of Depression in Adolescents: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2023 Nov 16;12:e48740. doi: 10.2196/48740. PMID 37971800

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Active Intervention | Usual Care
Started | 111 | 112
Completed | 96 | 98
Not Completed | 15 | 14

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Intervention | Usual Care | Total
Number analyzed (Participants) | 111 | 112 | 223
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 54 | 56 | 110
  Between 18 and 65 years | 57 | 56 | 113
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 17.3 (2.6) | 17.2 (2.7) | 17.3 (2.6)
Sex/Gender, Customized [Number; unit: participants]
  Gender Identity : Girl/Woman | 61 | 65 | 126
  Gender Identity : Boy/Man | 35 | 33 | 68
  Gender Identity : Non-binary | 13 | 16 | 29
  Gender Identity : Transgender | 13 | 10 | 23
  Gender Identity : Intersex | 1 | 0 | 1
  Gender Identity : Other | 8 | 4 | 12
  Gender Identity : I prefer not to say | 2 | 3 | 5
Sex: Female, Male [Count of Participants; unit: Participants] — Population: One participant from each group indicated that their sex at birth was "Unknown". Due to system constraints, it is not possible to enter anything other than Female or Male on this form.
  Participants
    number analyzed (Participants) | 110 | 111 | 221
    Female | 82 | 81 | 163
    Male | 28 | 30 | 58
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15 | 15 | 30
  Not Hispanic or Latino | 87 | 89 | 176
  Unknown or Not Reported | 9 | 8 | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 3
  Asian | 7 | 4 | 11
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 11 | 8 | 19
  White | 77 | 86 | 163
  More than one race | 11 | 11 | 22
  Unknown or Not Reported | 3 | 2 | 5
Patient Health Questionnaire-8 (PHQ-8) [Mean (Standard Deviation); unit: units on a scale] — The Patient Health Questionnaire (PHQ-8), an 8-item participant-report measure for screening for depression and for establishing depression severity. The total score, resulting from adding all item level scores, ranges from 0-24, with a higher score indicating greater depression symptom severity.
  units on a scale | 12.14 (4.28) | 12.59 (4.24) | 12.37 (4.26)

OUTCOME MEASURES:

1. Primary Outcome: Depressive Symptom Severity at Post-intervention
Description: Measured by the Patient Health Questionnaire (PHQ-8), an 8-item participant-report measure for screening for depression and for establishing depression severity. The total score ranges from 0-24, with a higher score indicating greater depression symptom severity.
Time Frame: Post-intervention (5 week timepoint)
Population: Intention to Treat
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Active Intervention | Usual Care
Number analyzed (Participants) | 111 | 112
units on a scale | 8.39 (0.38) | 11.03 (0.37)
Statistical Analysis 1: Comparison: Active Intervention vs Usual Care; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = -2.63, 95% CI 2-sided [-3.68 to -1.59], Standard Error of Mean 0.53

2. Secondary Outcome: Intervention Response at Post-intervention
Description: Measured by the Patient Health Questionnaire (PHQ-8) an 8-item participant-report measure for screening for depression and for establishing depression severity. The total score ranges from 0-24, with a higher score indicating greater depression symptom severity. Intervention response is defined as a 50% reduction in PHQ-8 score from baseline.
Time Frame: Change from baseline to post-intervention (5 weeks)
Population: Missing values imputed with multiple imputation.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Active Intervention | Usual Care
Number analyzed (Participants) | 111 | 112
percentage of participants
  Intervention Response (Yes) | 31.7 [22.5 to 40.8] | 11.6 [5.2 to 18.0]
  Intervention Response (No) | 68.3 [59.2 to 77.5] | 88.4 [82.0 to 94.8]
Statistical Analysis 1: Comparison: Active Intervention vs Usual Care; Missing values imputed with multiple imputation. P-values are obtained from a Pearson Chi-Squared test; differences and 95% CIs are obtained from a difference in proportions Z- test; Test type: Superiority; p < 0.001, Chi-squared; Difference in proportion z-test = 20.1, 95% CI 2-sided [9.1 to 31.0]

3. Secondary Outcome: Remission at Post-intervention
Description: Measured by the Patient Health Questionnaire (PHQ-8) an 8-item participant-report measure for screening for depression and for establishing depression severity. The total score ranges from 0-24, with a higher score indicating greater depression symptom severity. Remission is defined as a PHQ-8 score less than 5 at post-intervention.
Time Frame: Post-intervention (5 week timepoint)
Population: Missing values imputed with multiple imputation.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Active Intervention | Usual Care
Number analyzed (Participants) | 111 | 112
percentage of participants | 24.9 [16.4 to 33.4] | 9.4 [3.9 to 15.0]
Statistical Analysis 1: Comparison: Active Intervention vs Usual Care; P-values are obtained from a Pearson Chi-Squared test; differences and 95% CIs are obtained from a difference in proportions Z- test; Test type: Superiority; p = 0.003, Chi-squared; Difference in proportions z-test = 15.4, 95% CI 2-sided [5.3 to 25.6]

4. Secondary Outcome: Clinically-meaningful Reduction in Severity at Post-intervention
Description: Measured by the Patient Health Questionnaire (PHQ-8) an 8-item participant-report measure for screening for depression and for establishing depression severity. The total score ranges from 0-24, with a higher score indicating greater depression symptom severity. Clinically-meaningful reduction is defined as a ≥5 point reduction in PHQ-8 score from baseline.
Time Frame: Change from baseline to post-intervention (5 weeks)
Population: Intention to treat. Missing values are imputed with multiple imputation.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Active Intervention | Usual Care
Number analyzed (Participants) | 111 | 112
percentage of participants | 40.5 [30.9 to 50.1] | 15.8 [8.9 to 22.7]
Statistical Analysis 1: Comparison: Active Intervention vs Usual Care; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p < 0.001, Chi-squared; Difference in proportion z-test = 24.7, 95% CI 2-sided [13.0 to 36.4]

ADVERSE EVENTS:
Time Frame: Through study completion, up to 11 weeks after randomization
Arm/Group | Active Intervention | Usual Care
All-Cause Mortality (participants affected / at risk) | 0/111 | 0/112
Serious Adverse Events (participants affected / at risk) | 2/111 | 1/112
Other Adverse Events (participants affected / at risk) | 0/111 | 0/112
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Active Intervention (N=111) | Usual Care (N=112)
Hospitalization (Psychiatric disorders) | 2 | 0 — Hospitalization due to suicidal ideation or self-injurious behavior
Victim of violence (Social circumstances) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-01-24): https://cdn.clinicaltrials.gov/large-docs/52/NCT05462652/Prot_SAP_000.pdf